CLINICAL TRIAL: NCT03476902
Title: Feasibility, Acceptability, and Preliminary Efficacy of a Mobile App (nOCD) for OCD
Acronym: nOCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Helen Blair Simpson, Research Chief, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7572
Record Dates: First submitted 2018-03-12; First posted 2018-03-26 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: OCD; Mobile; Technology; CBT; Cognitive-Behavioral Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated Mobile Treatment (Experimental): Individuals will receive 4 introductory sessions with a therapist followed by weekly phone calls. Participants will utilize nOCD application to assist with treatment protocol adherence.
  Interventions: Behavioral: Therapist assisted mobile intervention

INTERVENTIONS:
Behavioral: Therapist assisted mobile intervention — Individuals will receive 4 introductory sessions with a therapist followed by weekly phone calls. Participants will utilize nOCD application to assist with treatment protocol adherence.

SUMMARY:
The purpose of this study is to evaluate the feasibility, acceptability, and potential usefulness of using a mobile application (nOCD) for treatment of obsessive compulsive disorder (OCD) in a sample of 25 adults (ages 18-65) in an 8 week trial. nOCD is a free iOS/Android application that provides treatment strategies. The study team will evaluate the effect of the application using gold-standard clinician-administered and self-report measures. Prior to downloading the application, participants will receive 4 (up to 5) in-person visit (orientation to the app and psychoeducation) and receive brief weekly phone check-ins. The long-term goal of this study is to use this information to develop new treatments for patients with OCD. All study procedures will be conducted on site at the New York State Psychiatric Institute.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility, acceptability, and potential usefulness of using a mobile app (nOCD) for treatment of OCD in a sample of 25 adults (ages 18-65). nOCD is a free iOS/Android app that provides EX/RP-consistent treatment strategies. The study team will evaluate the effect of the app using gold-standard clinician-administered and self-report measures. Prior to downloading the app, participants will receive 4 (up to 5) in-person visits and receive brief weekly phone check-in. The long term goal of this line of research is to increase access to evidence-based treatment and to ultimately reach more patients giving them access to tools to reduce their OCD symptoms and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-5 diagnosis of obsessive-compulsive disorder
* Age 18-65
* Not currently receiving psychotherapy focused on OCD symptoms, and no EX/RP within the past 12 weeks
* For those currently on medication: On a stable dose of psychiatric medication (for at least 12 weeks)
* Capacity to provide informed consent

Exclusion Criteria:

* Comorbid psychiatric conditions that significantly elevate the risk of study participation (e.g. psychotic disorders, bipolar disorder, evidence of dementia or other cognitive disorder, suicidality).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of using a therapist assisted mobile app using the System Usability Scale (SUS). | 8 weeks
  Feasibility and acceptability will be assessed using the System Usability Scale (SUS) at post treatment. SUS scores range from 0-100 with higher scores indicating better outcomes.
Effect of therapist assisted mobile app on OCD symptoms as assessed by the Yale-Brown Obsessive Compulsive Scale (Y-BOCS). | Baseline and approximately 8 weeks
  Reduction in OCD symptoms as assessed by the Yale-Brown Obsessive Compulsive Scale (Y-BOCS). Y-BOCS scores range from 0-40 with lower values representing better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Gershkovich, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gershkovich M, Middleton R, Hezel DM, Grimaldi S, Renna M, Basaraba C, Patel S, Simpson HB. Integrating Exposure and Response Prevention With a Mobile App to Treat Obsessive-Compulsive Disorder: Feasibility, Acceptability, and Preliminary Effects. Behav Ther. 2021 Mar;52(2):394-405. doi: 10.1016/j.beth.2020.05.001. Epub 2020 May 11. PMID 33622508
- See also: Center for OCD & Related Disorders Webpage — http://columbiapsychiatry.org/ocd